CLINICAL TRIAL: NCT01068717
Title: Bioequivalence Study of the Fixed Dose Combination of 2.5 mg Saxagliptin and 500 mg Metformin Tablet Relative to a 2.5 mg Saxagliptin (Onglyza) Tablet and a 500 mg Metformin (Glucophage Marketed in Canada by Sanofi-Aventis) Tablet Co-Administered to Healthy Subjects in the Fasted and Fed States
Brief Title: Bioequivalence Study of 2.5-mg Saxagliptin and 500-mg Glucophage in Tablets and a Fixed-dose Combination Tablet in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-118
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saxagliptin, 2.5 mg + Metformin, 500 mg (fasted state) (Other): Single oral doses of saxagliptin, 2.5 mg, and metformin, 500 mg, administered together as tablets in the fasted state
  Interventions: Drug: Saxagliptin, 2.5 mg + Metformin, 500 mg (fasted state)
- Saxagliptin, 2.5 mg/Metformin, 500 mg FDC (fasted state) (Other): Single oral dose of a 2.5-mg saxagliptin/500-mg metformin fixed-dose combination (FDC) tablet administered in the fasted state
  Interventions: Drug: Saxagliptin, 2.5 mg /Metformin, 500 mg FDC (fasted state)
- Saxagliptin, 2.5 mg + Metformin, 500 mg (fed state) (Other): Single oral doses of saxagliptin, 2.5 mg, and metformin, 500 mg, administered together as tablets in the fed state
  Interventions: Drug: Saxagliptin, 2.5 mg + Metformin, 500 mg (fed state)
- Saxagliptin, 2.5 mg/Metformin, 500 mg FDC (fed state) (Other): Single oral dose of saxagliptin, 2.5 mg/metformin, 500 mg, FDC tablet administered in the fed state
  Interventions: Drug: Saxagliptin, 2.5 mg /Metformin, 500 mg FDC (fed state)

INTERVENTIONS:
Drug: Saxagliptin, 2.5 mg + Metformin, 500 mg (fasted state) — Tablets, oral, 2.5-mg saxagliptin and 500-mg metformin, once daily, 1 week
  Other Names: Onglyza™; Glucophage™
  Arms: Saxagliptin, 2.5 mg + Metformin, 500 mg (fasted state)
Drug: Saxagliptin, 2.5 mg /Metformin, 500 mg FDC (fasted state) — Tablets, oral, 2.5-mg saxagliptin/500-mg metformin fixed-dose combination (FDC), once daily, 1 week
  Arms: Saxagliptin, 2.5 mg/Metformin, 500 mg FDC (fasted state)
Drug: Saxagliptin, 2.5 mg + Metformin, 500 mg (fed state) — Tablets, oral, 2.5-mg saxagliptin and 500-mg metformin, once daily, 1 week
  Other Names: Onglyza™; Glucophage™
  Arms: Saxagliptin, 2.5 mg + Metformin, 500 mg (fed state)
Drug: Saxagliptin, 2.5 mg /Metformin, 500 mg FDC (fed state) — Tablets, oral, 2.5-mg saxagliptin and 500-mg metformin FDC, once daily, 1 week
  Arms: Saxagliptin, 2.5 mg/Metformin, 500 mg FDC (fed state)

SUMMARY:
To demonstrate the bioequivalence of a 2.5-mg saxagliptin/500-mg metformin fixed-dose combination (FDC) tablet to that of 2.5-mg saxagliptin (Onglyza) and 500-mg metformin (Glucophage, marketed in Canada by Sanofi-Aventis) tablets coadministered to healthy participants in the fasted and fed states.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 55 years, inclusive
* Healthy participants as determined by a lack of clinically significant deviation from normal in medical history, physical examination, electrocardiograms, and clinical laboratory determinations
* Body Mass Index of 18 to 32 kg/m^2, inclusive

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of allergy to DPP-4 inhibitors or related compounds
* History of allergy or intolerance to metformin or other similar acting agents
* Previous exposure to saxagliptin
* Exposure to metformin within 3 months pervious to study drug administration
* Estimated creatinine clearance of <80 mL/min using the Cockcroft Gault formula

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled and randomly assigned to 1 of 4 treatment sequences: ADBC, BACD, CBDA, or DCAB. One participant withdrew from the study on Day -1 of Period 2 due to a family emergency and returned for early termination assessments on Day 4 of Period 2. She did not receive study drug in Period 2.
Groups:
- Treatment Schedule ADBC: (Treatment A) A single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment D) a single oral dose of 2.5-mg saxagliptin/500-mg metformin fixed-dose combination (FDC) in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment B) a single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment C) a single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fed state.
- Treatment Schedule BACD: (Treatment B) A single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment A) a single oral dose of saxagliptin 2.5-mg and metformin 500-mg tablets administered together in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment C) a single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fed state. Then, (Treatment D) a single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC administered in the fasted state.
- Treatment Schedule CBDA: (Treatment C) A single oral dose of saxagliptin 2.5-mg and metformin 500-mg tablets administered together in the fed state, followed by a 7-day (minimum) washout period. Then, (Treatment B) a single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC administered in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment D) a single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC administered in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment A) a single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fasted state.
- Treatment Schedule DCAB: (Treatment D) a single oral dose of 2.5-mg saxagliptin/500- mg metformin FDC administered in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment C) a single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fed state. Then, (Treatment A) a single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fasted state, followed by a 7-day (minimum) washout period. Then, (Treatment B) a single oral dose of 2.5-mg saxagliptin/500- mg metformin FDC administered in the fasted state.
Period: Period 1: Treatment Schedule Phase 1
Arm/Group | Treatment Schedule ADBC | Treatment Schedule BACD | Treatment Schedule CBDA | Treatment Schedule DCAB
Started | 7 | 6 | 7 | 7
Completed | 6 (Patient who withdrew returned for Treatment Periods 3 and 4.) | 6 | 7 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Patient withdrew; returned for period 3 | 1 | 0 | 0 | 0
Period: Period 2: Treatment Schedule Phase 2
Arm/Group | Treatment Schedule ADBC | Treatment Schedule BACD | Treatment Schedule CBDA | Treatment Schedule DCAB
Started | 6 | 6 | 7 | 7
Completed | 6 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3: Treatment Schedule Phase 3
Arm/Group | Treatment Schedule ADBC | Treatment Schedule BACD | Treatment Schedule CBDA | Treatment Schedule DCAB
Started | 7 (Patient who withdrew during Treatment Period 1 returned for Treatment Periods 3 and 4.) | 6 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 4: Treatment Schedule Phase 4
Arm/Group | Treatment Schedule ADBC | Treatment Schedule BACD | Treatment Schedule CBDA | Treatment Schedule DCAB
Started | 7 (Patient who withdrew during Treatment Period 1 returned for Treatment Periods 3 and 4.) | 6 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated: All participants who received study medication.
Arm/Group | All Treated
Number analyzed (Participants) | 27
Age, Customized [Mean (Standard Deviation); unit: years] | 33.6 (7.42)
Age, Customized [Median (Full Range); unit: Years] | 32 [23 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 5
  White | 22

OUTCOME MEASURES:

1. Primary Outcome: Observed Maximum Plasma Concentration (Cmax) of Saxagliptin, Tablets and Fixed-dose Combination (FDC), Administered to Participants in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: All participants who received at least 1 of the 4 treatments and had sufficient plasma concentration data to facilitate the calculation of at least 1 primary pharmacokinetic parameter for at least 1 of the treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: Saxagliptin and Metformin Tablets, Fasted: A single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fasted state, followed by a 7-day (minimum) washout period.
- Treatment B: Saxagliptin and Metformin FDC, Fasted: A single oral dose of 2.5-mg saxagliptin/500-mg metformin fixed-dose combination (FDC) administered in the fasted state, followed by a 7-day (minimum) washout period.
- Treatment C: Saxagliptin and Metformin Tablets, Fed: A single oral dose of saxagliptin 2.5-mg and metformin 500-mg tablets administered together in the morning within 5 minutes of completing a standard high-fat, high-calorie breakfast (fed state), followed by a 7-day (minimum) washout period.
- Treatment D: Saxagliptin and Metformin FDC, Fed: A single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC administered in the morning within 5 minutes of completing a standard high-fat, high-calorie breakfast (fed state), followed by a 7-day (minimum) washout period.
Arm/Group | Treatment A: Saxagliptin and Metformin Tablets, Fasted | Treatment B: Saxagliptin and Metformin FDC, Fasted | Treatment C: Saxagliptin and Metformin Tablets, Fed | Treatment D: Saxagliptin and Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
ng/mL | 10.54 (26) | 11.53 (26) | 12.71 (36) | 12.79 (37)
Statistical Analysis 1: Comparison: Treatment A: Saxagliptin and Metformin Tablets, Fasted vs Treatment B: Saxagliptin and Metformin FDC, Fasted; To demonstrate the bioequivalence of FDC tablet versus coadministration of saxagliptin and metformin tablets in the fasted and fed states, linear mixed model analyses were performed on log(Cmax), log[AUC(INF)], and log[AUC(0-T)] of saxagliptin and metformin, respectively. The factors in the model were sequence, period, and treatment as fixed effects and measurements within each subject as repeated measurements allowing for different covariance structures for the fasted and fed states; Test type: Non-Inferiority or Equivalence — Point estimates and 90% confidence intervals (CIs) were calculated for Treatment B to Treatment A and Treatment D to Treatment C ratios of geometric means for Cmax, AUC(INF), and AUC(0-T) of saxagliptin and metformin, respectively. Potency-corrected results were also provided. Bioequivalence will be concluded if the 90% CIs for the test-to-reference ratios of geometric means are entirely contained within 80% to 125% for both Cmax and AUC(INF). No adjustments were made for multiplicity; Ratio geometric least squares (LS) mean = 109.53, 90% CI 2-sided [102.67 to 116.85]
Statistical Analysis 2: Comparison: Treatment C: Saxagliptin and Metformin Tablets, Fed vs Treatment D: Saxagliptin and Metformin FDC, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 100.37, 90% CI 2-sided [85.70 to 117.56]

2. Primary Outcome: Observed Cmax of Metformin, Tablets and FDC, Administered to Participants in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Saxagliptin and Metformin Tablets, Fasted | Treatment B: Saxagliptin and Metformin FDC, Fasted | Treatment C: Saxagliptin and Metformin Tablets, Fed | Treatment D: Saxagliptin and Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
ng/mL | 1058.19 (23) | 1044.70 (25) | 810.08 (22) | 811.94 (20)
Statistical Analysis 1: Comparison: Treatment A: Saxagliptin and Metformin Tablets, Fasted vs Treatment B: Saxagliptin and Metformin FDC, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 99.02, 90% CI 2-sided [91.29 to 107.41]
Statistical Analysis 2: Comparison: Treatment C: Saxagliptin and Metformin Tablets, Fed vs Treatment D: Saxagliptin and Metformin FDC, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 100.21, 90% CI 2-sided [96.86 to 103.67]

3. Primary Outcome: Terminal Half-life (t1/2) of Saxagliptin and Metformin, Tablets and FDC, Administered to Participants in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Treatment A: Saxagliptin + Metformin Tablets, Fasted: A single oral dose of saxagliptin, 2.5-mg and metformin 500-mg tablets administered together in the fasted state, followed by a 7-day (minimum) washout period.
- Treatment B: Saxagliptin/Metformin FDC, Fasted: A single oral dose of 2.5-mg saxagliptin/500-mg metformin fixed-dose combination (FDC) administered in the fasted state, followed by a 7-day (minimum) washout period.
- Treatment C: Saxagliptin + Metformin Tablets, Fed: A single oral dose of saxagliptin 2.5-mg and metformin 500-mg tablets administered together in the morning within 5 minutes of completing a standard high-fat, high-calorie breakfast (fed state), followed by a 7-day (minimum) washout period.
- Treatment D: Saxagliptin/Metformin FDC, Fed: A single oral dose of 2.5-mg saxagliptin/500-mg metformin FDC administered in the morning within 5 minutes of completing a standard high-fat, high-calorie breakfast (fed state), followed by a 7-day (minimum) washout period.
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 25
Hours
  t1/2 saxagliptin | 6.16 (1.06) | 6.69 (0.90) | 5.99 (0.91) | 6.15 (0.79)
  t1/2 metformin | 11.05 (3.94) | 13.02 (5.37) | 10.72 (2.61) | 10.96 (4.03)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC[0-t]) for Saxagliptin, Tablets and FDC, Given in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Saxagliptin and Metformin Tablets, Fasted | Treatment B: Saxagliptin and Metformin FDC, Fasted | Treatment C: Saxagliptin and Metformin Tablets, Fed | Treatment D: Saxagliptin and Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
ng*h/mL | 50.28 (24) | 51.60 (23) | 59.00 (20) | 58.94 (19)
Statistical Analysis 1: Comparison: Treatment A: Saxagliptin and Metformin Tablets, Fasted vs Treatment B: Saxagliptin and Metformin FDC, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 102.34, 90% CI 2-sided [97.96 to 106.91]
Statistical Analysis 2: Comparison: Treatment C: Saxagliptin and Metformin Tablets, Fed vs Treatment D: Saxagliptin and Metformin FDC, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 99.78, 90% CI 2-sided [96.61 to 103.05]

5. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events, and Adverse Events (AEs) Leading to Discontinuation
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Continuously over Days 1 to 3 of treatment Periods 1, 2, 3, and 4
Population: All enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
Participants
  Death | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0
  AEs Leading to Discontinuation | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Hematology, Serum Chemistry, and Urinalysis Laboratory Test Results
Description: Clinically significant was determined by the investigator. Hematology tests included hemoglobin, hematocrit, red blood cell count, total leukocyte count (including differential), and platelet count. Serum chemistry tests included aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, lactate dehydrogenase, creatinine, blood urea nitrogen, uric acid, fasting glucose, total protein, albumin, sodium, potassium, chloride, calcium, phosphorus, and creatine kinase. Urinalysis included protein, glucose, blood, leukocyte esterase, specific gravity, and pH.
Time Frame: At screening visit, at Day -1 of Periods 1 through 4, and at discharge
Population: All enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
Participants
  Hematology test results | 0 | 0 | 0 | 0
  Serum chemistry test results | 0 | 0 | 0 | 0
  Urinalysis results | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Results
Description: Clinically significant was determined by the investigator. ECGs were recorded after participants had been supine for at least 5 minutes.
Time Frame: At screening visit, Day -1 of Period 1, and at study discharge
Population: All enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Body Temperature, Blood Pressure, or Heart Rate
Description: Clinically significant was determined by the investigator. Blood pressure and heart rate were measured after the participant had been seated quietly for at least 5 minutes.
Time Frame: At screening visit, prior to dosing on Day 1 of Periods 1 through 4, and at study discharge.
Population: All enrolled participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
Participants | 0 | 0 | 0 | 0

9. Primary Outcome: AUC[0-t] for Metformin, Tablets and FDC, Given in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Saxagliptin and Metformin Tablets, Fasted | Treatment B: Saxagliptin and Metformin FDC, Fasted | Treatment C: Saxagliptin and Metformin Tablets, Fed | Treatment D: Saxagliptin and Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
ng*h/mL | 8035.25 (22) | 7906.00 (21) | 7497.56 (23) | 7654.00 (19)
Statistical Analysis 1: Comparison: Treatment A: Saxagliptin and Metformin Tablets, Fasted vs Treatment B: Saxagliptin and Metformin FDC, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 102.34, 90% CI 2-sided [97.96 to 106.91]
Statistical Analysis 2: Comparison: Treatment C: Saxagliptin and Metformin Tablets, Fed vs Treatment D: Saxagliptin and Metformin FDC, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 101.82, 90% CI 2-sided [96.10 to 107.88]

10. Primary Outcome: AUC From Time 0 Extrapolated to Infinity (AUC[0-inf]) for Saxagliptin, Tablets and FDC, Given in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 26 | 26 | 25 | 25
ng*h/mL | 52.17 (24) | 53.73 (23) | 61.31 (20) | 60.88 (20)
Statistical Analysis 1: Comparison: Treatment A: Saxagliptin + Metformin Tablets, Fasted vs Treatment B: Saxagliptin/Metformin FDC, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (%) of geometric LS mean = 102.64, 90% CI 2-sided [98.31 to 107.16]
Statistical Analysis 2: Comparison: Treatment C: Saxagliptin + Metformin Tablets, Fed vs Treatment D: Saxagliptin/Metformin FDC, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (%) of geometric LS mean = 99.22, 90% CI [96.48 to 102.04]

11. Primary Outcome: AUC[0-inf] for Metformin, Tablets and FDC, Administered in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 26 | 26 | 25 | 25
ng*h/mL | 8142.68 (22) | 8070.25 (20) | 7612.94 (24) | 7690.69 (18)
Statistical Analysis 1: Comparison: Treatment A: Saxagliptin + Metformin Tablets, Fasted vs Treatment B: Saxagliptin/Metformin FDC, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 99.04, 95% CI 2-sided [92.90 to 105.59]
Statistical Analysis 2: Comparison: Treatment C: Saxagliptin + Metformin Tablets, Fed vs Treatment D: Saxagliptin/Metformin FDC, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio geometric LS mean = 102.77, 95% CI 2-sided [96.82 to 109.09]

12. Primary Outcome: Time to Achieve the Observed Maximum Plasma Concentration (Tmax) for Saxagliptin and Metformin, Tablets and FDC, Administered to Participants in the Fasted and Fed States
Time Frame: Days 1, 2, and 3 of Periods 1, 2, 3, and 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Saxagliptin + Metformin Tablets, Fasted | Treatment B: Saxagliptin/Metformin FDC, Fasted | Treatment C: Saxagliptin + Metformin Tablets, Fed | Treatment D: Saxagliptin/Metformin FDC, Fed
Number analyzed (Participants) | 27 | 26 | 26 | 26
Hours
  Tmax saxagliptin | 1.00 [0.25 to 3.00] | 0.75 [0.30 to 4.00] | 1.50 [0.50 to 8.00] | 1.00 [0.50 to 3.00]
  Tmax metformin | 3.00 [0.50 to 4.00] | 3.00 [1.00 to 6.00] | 4.00 [2.00 to 6.00] | 4.00 [1.50 to 8.00]

ADVERSE EVENTS:
Arm/Group | Fasted: 2.5mg Onglyza + 500mg Glucophage | Fasted: 2.5mg Saxa/500mg Metformin FDC | Fed: 2.5mg Onglyza + 500mg Glucophage | Fed: 2.5mg Saxa/500mg Metformin FDC
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 2/27 | 1/26 | 7/26 | 4/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted: 2.5mg Onglyza + 500mg Glucophage (N=27) | Fasted: 2.5mg Saxa/500mg Metformin FDC (N=26) | Fed: 2.5mg Onglyza + 500mg Glucophage (N=26) | Fed: 2.5mg Saxa/500mg Metformin FDC (N=26)
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Venipuncture site inflammation (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.